CLINICAL TRIAL: NCT03407794
Title: Effects of Fermented Vegetables on Markers of Inflammation and Composition of the Intestinal Microflora in Overweight and Obese Women
Brief Title: Effects of Fermented Vegetables on Gut Microflora and Inflammation in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Florida (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Principal Investigator, Andrea Arikawa, Assistant Professor, University of North Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10334264-2
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-11

CONDITIONS: Inflammation; Women's Health; Gastrointestinal Microbiome
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: This is a randomized parallel-arm trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study investigators will be blinded to the treatment conditions and the outcome assessors will only have access to study ID numbers when conducting the lab analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants randomized into the control group will be asked to follow their usual diet during the 6 weeks of the intervention.
- Fermented vegetable (Experimental): Participants randomized into the fermented vegetable group will receive 1/2 cup per day of fermented vegetables, including cabbage, carrots or pickles, for 6 weeks.
  Interventions: Other: Fermented vegetable
- Non-fermented vegetable (Active Comparator): Participants randomized into the non-fermented vegetable group will receive 1/2 cup per day of non-fermented vegetables, including cabbage, carrots or pickles, for 6 weeks.
  Interventions: Other: Non-fermented vegetable

INTERVENTIONS:
Other: Fermented vegetable — The intervention is to consume 1/2 cup fermented vegetables every day for 6 weeks
  Arms: Fermented vegetable
Other: Non-fermented vegetable — The intervention is to consume 1/2 cup of non-fermented vegetables every day for 6 weeks
  Arms: Non-fermented vegetable

SUMMARY:
This proposal will examine whether daily consumption of fermented vegetables for 6 weeks can impact the gut microflora and markers of inflammation of women between the ages of 18-70 years.

DETAILED DESCRIPTION:
Interested participants will be invited to an orientation where study procedures will be explained in detail. Once the consent form is signed participants will schedule a visit to provide blood, urine and stool samples at the beginning of the intervention at which point they will be randomized into one of three groups: a fermented vegetable group (1/2 cup per day for 6 weeks), a non-fermented vegetable group (1/2 cup per day for 6 weeks) and a control group (usual diet). Both vegetable groups will receive weekly deliveries of the vegetables to be consumed. Following 6 weeks, participants will provide blood, urine and stool samples one more time. Participants will also fill out questionnaires related to dietary intake, demographics, physical activity, prescription medication use and gastrointestinal function. Compliance will be monitored weekly via a gastrointestinal function log where participants will be asked to enter whether they consumed or not the vegetable provided each day, as well as any side effects of consumption.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18.5-40 kg/m2
* Non-smoker
* No previous diagnosis of cancer
* No thyroid disease
* No diabetes
* Willing to consume 1/2 cup of vegetables daily for 6 weeks
* No use of psychotic or depression medication
* No medication to lose weight
* Not on a weight loss diet
* No use of antibiotics over the past 3 months
* No consumption of fermented vegetables on a regular basis
* No history of autoimmune disease, including gastrointestinal disease

Exclusion Criteria:

* BMI <18.5 or >40 kg/m2
* Smoker
* Taking medications that affect appetite or body weight
* Uncontrolled Hypertension
* Diabetes
* Not willing to consume 1/2 cup of vegetables daily for 6 weeks
* Willing to show up at two appointments
* Following a fad diet
* Using antibiotics frequently
* Diagnosed with autoimmune disease, like psoriasis, rheumatoid arthritis, thyroid disease, colitis
* Regular consumption of fermented vegetables

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Enrollment: 34 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan at the moment.

REFERENCES:
- [Background] Kim EK, An SY, Lee MS, Kim TH, Lee HK, Hwang WS, Choe SJ, Kim TY, Han SJ, Kim HJ, Kim DJ, Lee KW. Fermented kimchi reduces body weight and improves metabolic parameters in overweight and obese patients. Nutr Res. 2011 Jun;31(6):436-43. doi: 10.1016/j.nutres.2011.05.011. PMID 21745625
- [Background] Han K, Bose S, Wang JH, Kim BS, Kim MJ, Kim EJ, Kim H. Contrasting effects of fresh and fermented kimchi consumption on gut microbiota composition and gene expression related to metabolic syndrome in obese Korean women. Mol Nutr Food Res. 2015 May;59(5):1004-8. doi: 10.1002/mnfr.201400780. Epub 2015 Mar 23. PMID 25688926

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Fermented Vegetable | Non-fermented Vegetable
Started | 10 | 11 | 13
Completed | 10 | 10 | 11
Not Completed | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Fermented Vegetable | Non-fermented Vegetable | Total
Number analyzed (Participants) | 10 | 11 | 13 | 34
Age, Continuous [Median (Full Range); unit: years] | 27.5 [21 to 50] | 37 [19 to 63] | 44 [18 to 69] | 37 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 13 | 34
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 8 | 9 | 12 | 29
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 6 | 8 | 10 | 24
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 13 | 34
Education: Some college, College degree, Graduate degree [Count of Participants; unit: Participants]
  Some College | 2 | 3 | 1 | 6
  College Degree | 5 | 3 | 6 | 14
  Graduate Degree | 3 | 5 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: C-reactive Protein
Description: Marker of systemic inflammation: serum CRP
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Control | Fermented Vegetable | Non-fermented Vegetable
Number analyzed (Participants) | 10 | 11 | 10
ng/mL | 160.7 [0 to 746] | 173.4 [0 to 375] | 211.4 [0 to 228]

2. Primary Outcome: Shannon Index
Description: The Shannon Index is a measure of diversity of microbial species that takes into account both abundance (the number of species present) and evenness (how close the numbers for each species are). The Shannon index can be calculated using the following equation: H= -∑(i=1)^s pi ln(pi). A value of zero for H indicates that a community has only one species. The higher the value of H, the higher the diversity of species in a particular community.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: Shannon index
Arm/Group | Control | Fermented Vegetable | Non-fermented Vegetable
Number analyzed (Participants) | 9 | 10 | 11
Shannon index | 3.14 [3.0 to 3.5] | 3.34 [3.3 to 3.7] | 3.38 [3.2 to 3.58]

3. Secondary Outcome: BMI
Description: Measured using a multifrequency bioimpedance scale
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: kg/m2
Arm/Group | Control | Fermented Vegetable | Non-fermented Vegetable
Number analyzed (Participants) | 10 | 10 | 11
kg/m2 | 22.8 [22 to 28] | 23.3 [22 to 28] | 26.7 [22.5 to 27.2]

4. Secondary Outcome: Body Fat Percentage
Description: Measured using a multifrequency bioimpedance scale
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: % body fat
Arm/Group | Control | Fermented Vegetable | Non-fermented Vegetable
Number analyzed (Participants) | 10 | 10 | 11
% body fat | 31.1 [25 to 35.5] | 31.4 [22 to 41] | 36.8 [34.8 to 39.5]

5. Secondary Outcome: Systolic Blood Pressure
Description: Measured using an electronic blood pressure cuff
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Control | Fermented Vegetable | Non-fermented Vegetable
Number analyzed (Participants) | 10 | 10 | 11
mmHg | 104 [89 to 111] | 121 [108 to 122] | 107 [104 to 121]

6. Secondary Outcome: Lipopolysaccharide
Description: Marker of inflammation in serum
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: micrograms/mL
Arm/Group | Control | Fermented Vegetable | Non-fermented Vegetable
Number analyzed (Participants) | 10 | 10 | 11
micrograms/mL | 12.7 [8.1 to 14.9] | 12.7 [10.5 to 16.5] | 13 [11 to 15.5]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: All study participants were healthy and no serious adverse events were expected.
Arm/Group | Control | Fermented Vegetable | Non-fermented Vegetable
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 3/10 | 6/10 | 9/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=10) | Fermented Vegetable (N=10) | Non-fermented Vegetable (N=11)
Bloating (Gastrointestinal disorders) | 0 (0) | 5 (20) | 6 (17)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (3)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Abdominal Pail (Gastrointestinal disorders) | 1 (10) | 1 (4) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
This was a small pilot and feasibility study. There were few subjects in each group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT03407794/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT03407794/ICF_001.pdf